CLINICAL TRIAL: NCT03249519
Title: Multimodal Therapy of Advanced Cervical Cancer With Radiotherapy or Chemoradiation, Interstitial Brachytherapy in Combination With Hyperthermia
Brief Title: Radiation Therapy or Chemoradiation, Interstitial Brachytherapy in Combination With Hyperthermia in Advanced Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HyZer_RCT_IBT
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Cervical Cancer
Keywords: Radiation therapy; Chemoradiation; Brachytherapy; Hyperthermia; Cervical cancer; Multimodality treatment of advanced cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Hyperthermia | interventions — Radiation; Radiotherapy; Brachytherapy; Cisplatin; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard Arm (Experimental): Radiation therapy: 50.4 Gy Brachytherapy: 35-40 Gy Chemotherapy: Cisplatin weekly 40mg/m^2 (6 cycles) Hyperthermia: 10 times
  Interventions: Radiation: Radiation; Radiation: brachytherapy; Drug: Cisplatin; Other: Hyperthermia

INTERVENTIONS:
Radiation: Radiation — 50.4 Gy
  Other Names: Radiation therapy
Radiation: brachytherapy — 35-40 Gy
  Other Names: Interstitial brachytherapy
Drug: Cisplatin — weekly 40 mg/m^2 (6cycles)
Other: Hyperthermia — 10 times

SUMMARY:
The combination of radiation therapy or chemoradiation with Interstitial brachytherapy for advanced cervical cancer (pN+, FIGO-Stage II B - IV A is standard of therapy. The radio- and chemosensitive effect of an additional hyperthermia might improve the clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed carcinoma of the Cervix
* FIGO-Stage IIB-IVA; earlier stages when inoperable or according to patient's wish
* clinical M0; except: involvement of para-aortic lymph nodes
* Age ≥ 18 years
* ECOG ≤ 2
* Informed consent of the patient

Exclusion Criteria:

* Pre-existing uncontrolled cardiac disease, signs of cardiac failure, or rhythm disturbances requiring therapy
* Cardiac Pacemaker
* Myocardial infarction within the past 12 months
* Congestive heart failure
* Complete bundle branch block
* New York Heart Association (NYHA) class III or IV heart disease
* Disease that would preclude chemoradiation or deep regional hyperthermia
* Metal implants (length > 2cm or dense clusters of marker clips in the pelvis)
* Active or therapy-resistent bladder infections
* Pre-existing or concommitant immunodeficiency Syndrome
* Pregnant or lactating women
* Patients not willing to use effective contraception during and up to 6 months after therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 999 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2094-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Disease free survival (local / distant / overall) | 5 years
Safety by Toxicity assessment according to NCI CTCAE v4.0 | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Erlangen, Strahlenklinik, Erlangen, Germany